CLINICAL TRIAL: NCT06393972
Title: The Efficacy and Safety of Tofacitinib in Patients With Glucocorticoid Resistant ICIs-related Myocarditis: a Single-arm, Prospective, Phase 2 Trial
Brief Title: The Efficacy and Safety of Tofacitinib in Patients With Glucocorticoid Resistant ICIs-related Myocarditis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Tianshu Liu, Clinical Professor, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSLCYJ202353
Record Dates: First submitted 2023-11-23; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Glucocorticoid Resistant ICIs-related Myocarditis
MeSH Terms: interventions — tofacitinib; BID protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tofacitinib (Experimental): Tofacitinib in patients with glucocorticoid resistant ICIs-related myocarditis
  Interventions: Drug: Tofacitinib 5 MG BID

INTERVENTIONS:
Drug: Tofacitinib 5 MG BID — Tofacitinib 5 MG BID

SUMMARY:
The efficacy and safety of Tofacitinib in patients with glucocorticoid resistant ICIs-related myocarditis: a single-arm, prospective, phase 2 trial

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Patients treated with ICI immunotherapy (monotherapy or combination), including anti-PD1, anti-PDL1, anti-CTLA4; and including any type of cancer (even those in which ICI is not currently approved by regulatory)
3. Definite, probable or possible ICI-induced myocarditis according to the diagnostic criteria of the most recent expert consensus recommendations (e.g27, to be updated with any new recommendations to be published)
4. corticosteroid-resistant ICI-myocarditis: Corticosteroid-resistant ICI-myocarditis is defined by the absence of decrease in troponin levels or the appearance/persistence of severity criteria despite receiving prednisone dose ≥0.5 mg/kg/day for ≥2 days.
5. Signature of informed consent before any trial procedure from the patient or legal representative or the close relative
6. Patients covered by social security regimen (excepting AME)
7. Withhold of ICI

Exclusion Criteria:

1. Untreated and/or uncontrolled bacterial, fungal, or viral infection Pregnancy, breast-feeding or planning to become pregnant during the study period
2. For women of childbearing age, lack of effective contraception throughout the duration of participation in the study
3. Being treated with tofacitinib within 3 months prior to inclusion Known hypersensitivity to abatacept or belatacept
4. Being treated with anti-thymoglobulin, or alemtuzumab within 6 weeks of the first scheduled dose of abatacept
5. Patient participating to another interventional study (RIPH 1 only) People under legal protection measure (tutorship, curatorship or safeguard measures)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality within three months | The first three months after tofacitinib administration
  All-cause mortality within three months

SECONDARY OUTCOMES:
All-cause mortality within six months | The firs six months after tofacitinib administration
  All-cause mortality within six months
Progression-free survival | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Progression-free survival
Overall survival | From date of enrollment until the date of death from any cause, assessed up to 24 months"
  Overall survival
Safety and tolerability based on incidence of treatment-emergent adverse events | through study completion, an average of 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0